CLINICAL TRIAL: NCT04866927
Title: Use of Stable Isotopic Dilution to Assess Protein Digestibility From Fava Bean and to Evaluate Amino Acid Bioavailability
Brief Title: Bioavailability of Proteins From Plant Based Diets
Status: Completed | Type: Observational
Sponsor: International Atomic Energy Agency (Other Government)
Collaborators: AgroParisTech (Other); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Centre National De L'énergie, Des Sciences Et Techniques Nucléaires (Other Government)
Responsible Party: Principal Investigator, Khayour Meriam, Principal investigator, International Atomic Energy Agency
Other Study IDs: E43031
Record Dates: First submitted 2021-04-16; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Protein Malabsorption; Nutritional Deficiency; Nutritional Stunting
Keywords: Proteins; Digestibility; Bioavailability; Indispensable Amino Acids; Plant-based food; Plant diet; Nutrition; Food security; Fava Bean; Vegetal proteins
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults: Inclusion criteria: Healthy, non-pregnant women, adults aged 18-65 years, not taking any medication, including NSAIDs, not taking antibiotics within 4 weeks of study, BMI within 18-35 range.
  Exclusion criteria: Children and elderly (over 65), pregnant women, individuals diagnosed with non-communicable or communicable disease, being under restrictive diet, antibiotics within 4 weeks of study, medications within 4 weeks of study.
  Interventions: Dietary Supplement: Use of stable isotopic dilution to assess protein digestibility from Faba bean and to evaluate amino acid bioavailability

INTERVENTIONS:
Dietary Supplement: Use of stable isotopic dilution to assess protein digestibility from Faba bean and to evaluate amino acid bioavailability — Each participant will receive a test meal containing 13C labelled spirulina, 2H labelled Fava bean and 13C phenylalanine. The test meal will be divided on 11 subdoses: 3 sub-doses will be administrated at T0 and 1 subdose will be administrated at 1, 2, 3, 4, 5, 6 and 7h. The remaining sub-dose will be kept for measurement of IAA in the test meal. After eating the test meal, blood, urine and breath samples will be collected from each participant at the baseline (T0) and after 5-6, 7h and 8h.

SUMMARY:
Proteins play an important role as structural and functional components for the human body and prevent stunting. Protein quality has a great importance in meeting the nutritional needs of populations across the world throughout the life course, particularly during pregnancy and early childhood. Dietary protein deficiency is mainly due to protein indigestibility limiting indispensable amino acids (IAAs) bioavailability. In Morocco, as it's the case in many developing countries, diet is mainly based on a large consumption of cereals, fruits, vegetables and pulses, and is generally low in meat, which is the main source of protein and IAA.

The general objective of this study is to evaluate the digestibility of Fava bean proteins and bioavailability of IAA using a dual-tracer method with stable isotopes.

DETAILED DESCRIPTION:
This study aims to develop stable isotope labeled protein of bean cultures that could be used for other local common foods, to quantify dietary indispensable amino acids from beans made available to the body for optimal growth, development and function and to participate in the development of a simple method to assess protein quality in vulnerable populations.

The project is divided in two parts: the first part of harvesting and production of deuterium labeled fava beans. The optimization test done the first year has shown that the best protocol for labelling was a pulse with 25% D2O followed with subsequent labeling with 2.5% D2O during 20 days.

The second part is the intervention stuy that is going to be conducted on 6 healthy volunteers (3 males, 3 females). Each participant will receive a test meal containing 13C labelled spirulina, 2H labelled Fava bean and 13C phenylalanine. The test meal will be divided on 11 subdoses: 3 sub-doses will be administrated at T0 and 1 subdose will be administrated at 1, 2, 3, 4, 5, 6 and 7h. The remaining sub-dose will be kept for measurement of IAA in the test meal. After eating the test meal, blood, urine and breath samples will be collected from each participant at the baseline (T0) and after 5-6, 7h and 8h.

ELIGIBILITY:
Inclusion Criteria:

Healthy, non-pregnant adults 18-65 years of age

Not taking any medication, including NSAIDs Not taking antibiotics within 4 weeks of study BMI within 18-35 range Stable weight

Exclusion Criteria:

Children and elderly (over 65)

Pregnancy Diagnosed with non-communicable or communicable disease Being under restrictive diet Antibiotics within 4 weeks of study Medications within 4 weeks of study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals who fit in the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Relative Amino Acid Digestibility | One year
  The digestibility of each IAA from the 13C-labeled spirulina protein and TCF is an IAA-specific term used to correct for loss of a 2H atom during transamination.
DIAAS | One year
  The digestible indispensable amino acid score (DIAAS), representing the content of each IAA, along with the digestibility of each IAA, in relation to the human requirement pattern was also calculated.

SECONDARY OUTCOMES:
Scientific articles | By the end of 2020
  Publication of scientific reports and peer-reviewed papers and conference presentations.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed El Mzibri, Principal Investigator — Head of the Division of Life Sciences - CNESTEN; Hassan Aguenaou, Study Director — Director of Nutrition RDC of Morocco
Locations (1):
- Joint Research Unit in Nutrition and Food, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khayour M, Benmhimdane A, Calvez J, Saeid N, Khodorova N, Belghiti H, El Hamdouchi A, El Kari K, Owino V, Tome D, Aguenaou H, Mentag R, El Mzibri M, Gaudichon C. Indispensable Amino Acid Digestibility of Moroccan Fava Bean Using the Dual Isotope Method in Healthy Adults. J Nutr. 2023 Feb;153(2):451-458. doi: 10.1016/j.tjnut.2022.11.015. Epub 2022 Dec 24. PMID 36894238